CLINICAL TRIAL: NCT02300376
Title: Designing a Bayesian Model of the Plasma Clearance of Calcium Edetate de Sodium, With a Limited Sampling Strategy for the Calculation of Glomerular Filtration Rate (GFR) and Validity Assessment Compared to the Renal Clearance of Inulin : DFGBay
Brief Title: Designing a Bayesian Model of the Plasma Clearance of Calcium Edetate de Sodium for the Calculation of GFR and Validity Compared to the Renal Clearance of Inulin
Acronym: DFGBay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I13034
Record Dates: First submitted 2014-10-28; First posted 2014-11-25 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2016-06

CONDITIONS: Kidney Disease
Keywords: GFR; Bayesian model; plasma clearance; Calcium edetate de sodium; Inulin
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium edetate de sodium versus inulin (Experimental): The designing a Bayesian model of the plasma clearance of Calcium edetate de sodium is compared to the renal clearance of Inulin.
  Interventions: Drug: Dosage of Calcium edetate de sodium

INTERVENTIONS:
Drug: Dosage of Calcium edetate de sodium — There is no medical data for the use of Calcium edetate de sodium as a tracer to assess GFR. Calcium edetate de sodium is a treatment for lead intoxication. The extension of use as a tracer comes from its exclusive elimination by glomerular filtration. Plasma and renal clearance of Calcium edetate de sodium and Inulin will be measured for every included patient during a hospital day care (V1). For transplanted patients, plasma clearance of Calcium edetate de sodium will be repeated within one week (more or less 48hours) during annual medical check-up of renal transplantation.

SUMMARY:
Diagnosis of patients with renal insufficiency and recommendations for medical treatment of patients who suffer from chronic renal failure are based on the different stages of Glomerular Filtration Rate (GFR). Many formulas exist to assess GFR. However these formulas are unreliable in many clinical situations (old people, obese patients…). Methods for measuring GFR using exogenous tracers exist: Inulin and 51Cr-EDTA are historical reference tracers. Renal clearance of Inulin is the gold standard. However, using these methods is restricted to specialized services because it is long and expensive.

There is no medical data for the use of Calcium edetate de sodium as a tracer to assess GFR. Calcium edetate de sodium is a treatment for lead intoxication. The extension of use as a tracer comes from its exclusive elimination by glomerular filtration.

Plasma and renal clearance of Calcium edetate de sodium and Inulin will be measured for every included patient during a hospital day care (First visit V1). For transplanted patients, plasma clearance of Calcium edetate de sodium will be repeated within one week (more or less 48hours) during annual medical check-up of renal transplantation (Second visit V2).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for V1:
* For transplanted patients : patients from 18 to 80 years, after estimation of their renal function by MDRDs formulas (MDRD = Modification of Diet in Renal Disease) , regardless their nephropathy, regardless the age of the transplantation, with a normal state body hydratation, with a social insurance and who have given their prior consent.
* For other patients : patients from 18 to 80 years, after estimation of their renal function by MDRDs formulas, who need a reliable assess of their renal function, with a normal state body hydratation, with a social insurance and who have given their prior consent.
* Inclusion criteria for V2: Transplanted patients who have participated to V1, with stable clinical conditions, with a stable GFR (less than 30% variation of creatinine clearance by MDRDs formulas) and who have given their prior consent.

Exclusion Criteria:

* Hypersensitivity to Calcium edetate de sodium
* Inulin or excipients
* Lead or other heavy metal intoxication
* Volume expansion or dehydration
* Acute renal disease
* Bladder voiding affections
* Coagulation disorders
* Poor venous capital
* People in guardianship
* Patients already involved in an other research
* Women in child bearing age without any method of contraception
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To estimate the DFG by the Bayesian model | 1 week
  the DFG assessed by the Bayesian model of the plasma clearance of Calcium edetate de sodium.

SECONDARY OUTCOMES:
Concordance of GFRBay | 1 week
  Concordance of the Bayesian model of GFR measured during V1 and during V2 to determine the reliability of the method

CONTACTS AND LOCATIONS:
Overall Officials: Julien ALLARD, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- University Hospital, Limoges, France